CLINICAL TRIAL: NCT01758003
Title: Patterns of Physical Activity in a Healthy Population Aged Over 40 Years Old
Brief Title: Physical Activity in Healthy Over 40s
Status: Completed | Type: Observational
Sponsor: University of Ulster (Other)
Responsible Party: Principal Investigator, Judy Bradley, Professor of Physiotherapy, University of Ulster
Other Study IDs: 12/08
Record Dates: First submitted 2012-12-22; First posted 2012-12-31 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Physical Activity
Keywords: Physical Activity; Sedentary Behaviour; Healthy Volunteer; Quality of Life; Exercise Capacity; Transtheoretical Model
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary aim of this research is to examine physical activity in a healthy population aged over 40 years old.

Subsidiary aims of this research are:

1. To establish normative values for physical activity levels, exercise capacity, quality of life and readiness to change physical activity behaviour (stages of change, self-efficacy, decisional balance and processes of change) in a healthy population age-matched to a population with bronchiectasis.
2. To explore physical activity levels, exercise capacity and quality of life in a healthy population age-matched to a population with bronchiectasis.
3. To explore readiness to change physical activity behaviour (stages of change, self-efficacy, processes of change and decisional balance) in a healthy population compared to a population with bronchiectasis.

DETAILED DESCRIPTION:
The current study is running alongside an externally funded project measuring physical activity levels in patients with bronchiectasis (ClinicalTrials.gov ID: NCT01569009). In order to more fully understand physical activity behaviours in bronchiectasis, it is important to compare the patterns of physical activity, exercise capacity and quality of life of the patients with bronchiectasis to a healthy age-matched population.

For a healthy population of similar age to patients with bronchiectasis, little applicable research currently exists with regard to normative values of physical activity and sedentary behaviour. In this particular study, we will measure physical activity levels in healthy individuals age-matched to patients with bronchiectasis. The most commonly used questionnaire to assess physical activity is the International Physical Activity Questionnaire. Pedometers are inexpensive devices which can be used to assess daily step count and time spent in walking. Activity monitors are more expensive and require technical expertise for analysis and interpretation. However, they provide more in-depth information on pattern, quantity and intensity of activity including daily sedentary time. In this study, the investigators will use the ActiGraph activity monitor, ActivPAL activity monitor, DigiWalker pedometer and IPAQ to measure the physical activity levels in healthy individuals age-matched to patients with bronchiectasis. This study will not focus on participants who engage in high levels of physical activity as they are unlikely to represent the physical activity levels of patients with bronchiectasis.

This study will include the Modified Shuttle Test. Exercise capacity measured by the Modified Shuttle Test is normally only utilized in respiratory disease populations such as patients with cystic fibrosis. However, it has recently been highlighted that there is a need for reference data in healthy populations. This study will also use the EQ-5D-5L questionnaire to assess quality of life. Preliminary testing of the EQ-5D-5L questionnaire, an update to the well-researched EQ-5D-3L, has only recently been conducted. There is a need for studies to provide more normative data on the EQ-5D-5L.

This study will also assess readiness to change physical activity behaviour in a healthy population utilising transtheoretical model components such as stages of change, self-efficacy, decisional balance and processes of change; which have all been shown to be important in physical activity behaviour. Understanding healthy individuals' perspectives on readiness to change physical activity behaviour and the links between important outcomes will help to inform future physical activity interventions.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 40 years
* does not participate in regular exercise or participates in regular exercise at a moderate level ≤ 3 hours/week
* ≤ 10 pack-year history of smoking
* does not suffer from any concomitant condition which may prevent participation in physical activity
* answered 'No' to all questions in the Medical Questionnaire

Exclusion Criteria:

* participates in regular exercise at a moderate level > 3 hours/week
* pregnancy
* any concomitant condition which may prevent participation in physical activity
* answered 'Yes' to any questions in the Medical Questionnaire

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy convenience sample
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Step counts measured by the ActiGraph GT3X+ activity monitor | Seven days
  Participants will wear the ActiGraph GT3X+ activity monitor for seven consecutive full days between Visit 1 (Day 0) and Visit 2 (Day 8).

SECONDARY OUTCOMES:
Step counts measured by the ActivPAL activity monitor | Seven days
  Participants will wear the ActivPAL activity monitor for seven consecutive full days between Visit 1 (Day 0) and Visit 2 (Day 8).
Number of steps measured by the Yamax CW-700 DigiWalker pedometer | Seven days
  Participants will wear the Yamax CW-700 DigiWalker pedometer for seven consecutive full days between Visit 1 (Day 0) and Visit 2 (Day 8).
Physical activity levels and sitting time using the International Physical Activity Questionnaire | Day 8
  Participants will complete the International Physical Activity Questionnaire at Visit 2 (Day 8). It will be used to measure participants' time spent in physical activity in the last seven days and also to provide self-reported sitting time.
Quality of Life using the EuroQOL-5D-5L | Day 8
  Participants will complete the EuroQOL-5D-5L at Visit 2 (Day 8).
Stage of change in terms of physical activity using the Stages of Change Questionnaire | Day 8
  Participants will complete the Stages of Change Questionnaire at Visit 2 (Day 8). The Stages of Change Questionnaire is the temporal part of the transtheoretical model. It will be used to determine the current stage of change the participant is at in terms of their physical activity behaviour.
Confidence to undertake physical activity using Marcus's Self-Efficacy Questionnaire | Day 8
  Participants will complete Marcus's Self-Efficacy Questionnaire at Visit 2 (Day 8). Marcus's Self-Efficacy Questionnaire is a component of the transtheoretical model. It will provide more detailed information on each individual's confidence to undertake physical activity in different situations.
Perception of the benefits and negative aspects of physical activity using Marcus's Decisional Balance Questionnaire | Day 8
  Participants will complete Marcus's Decisional Balance Questionnaire at Visit 2 (Day 8). Marcus's Decisional Balance Questionnaire is a component of the transtheoretical model. It will assess each individual's perceptions of the benefits and negative aspects of physical activity.
Strategies used to progress through the different stages of change using Marcus's Processes of Change Questionnaire | Day 8
  Participants will complete Marcus's Processes of Change Questionnaire at Visit 2 (Day 8). Marcus's Processes of Change Questionnaire is a component of the transtheoretical model. It describes the strategies and techniques individuals use to progress through the different stages of change.
Perception of the feasibility and acceptability of the physical activity outcome measures | Day 8
  The researcher and the participants will answer the feasibility and acceptability questions at Visit 2 (Day 8). The feasibility and acceptibility questions were designed for this study to assess the researchers' and participants' perspectives of the feasibility and acceptability of the physical activity outcome measures (ActiGraph, ActivPAL, pedometer and International Physical Activity Questionnaire.
Exercise Capacity using the Modified Shuttle Test | Day 8
  Participants will complete the Modified Shuttle Test at Visit 2 (Day 8).

CONTACTS AND LOCATIONS:
Overall Officials: Judy Bradley, PhD, Principal Investigator — University of Ulster
Locations (1):
- University of Ulster, Jordanstown, Antrim, United Kingdom